CLINICAL TRIAL: NCT03804047
Title: KITAMS: Kinesio Tape and Physical Function in Persons With Multiples Sclerosis
Acronym: KITAMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern Illinois University (Other)
Responsible Party: Principal Investigator, Emerson Sebastião, Assistant Professor, Northern Illinois University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS18-0012
Record Dates: First submitted 2019-01-10; First posted 2019-01-15 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Multiple Sclerosis
Keywords: Kinesio Tape; Physical functioning; Disability
MeSH Terms: conditions — Multiple Sclerosis | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: Two arm randomized controlled trial (Pre; Post)
Who Masked: Participant
Masking Description: Randomization will done using concealed allocation with the use of opaque envelopes. Envelopes will be spread out over a table and participants will choose one to give it to the Physical Therapist (PT). The PT will open the envelope to check the type of tape (without showing or saying it to the participant) to be applied (kinesio or Sham tape). Participants are unaware about tape categorization "treatment" or "placebo" as the tapes are unlabeled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Tape (KTG) (Experimental): Participants allocated into the KTG will receive a single time application of the kinesio tape flexible tape (Kinesio® Tex, Albuquerque, NM, USA) in the upper-body (i.e., back part of the trunk) and in the lower-body (i.e., legs and ankle) according to standardized procedures (https://kinesiotaping.com/how-to/). The tape is latex-free and wearable for weeks without causing skin irritation (i.e., hypoallergenic); and safe for populations ranging from pediatric to geriatric. The tape will be applied by a Physical Therapist with experience in tape application. Tape application will be conducted in a private room with a complete structure for the procedure.
  Interventions: Other: kinesio tape
- Sham Tape (STG) (Sham Comparator): Participants allocated into the STG will receive a single time application of an inflexible tape (i.e., sham tape) in the same body segments as the intervention condition. Tape application will be conducted in a private room with a complete structure for the procedure.
  Interventions: Other: kinesio tape

INTERVENTIONS:
Other: kinesio tape — kinesio tape is a therapeutic method used in the treatment of various musculoskeletal and neuromuscular deficits to provide support for muscles and increase or inhibit muscle recruitment, to correct joint malalignment, decrease swelling, and pain relieve

SUMMARY:
Multiple sclerosis (MS) is a disease that causes damage within the central nervous system and results in deficits of body functions. The investigators propose a pilot randomized controlled trial examining the acute effect of kinesio tape application in various body segments on balance, mobility, physical functioning, and pain in persons with MS (pwMS) aged 18 to 55 years old. The investigators will objectively assess balance using a force platform and mobility and physical functioning will be assessed using standardized tests (i.e., Timed Up and Go, Timed 25-foot Walk, 6-minute Step Test, Six Spot Step Test). The trial will recruit 24 pwMS aged 18 to 55 years with mild-to-moderate MS-related disability who will be randomized into intervention (Kinesio Tape) or control conditions (Sham/Inflexible Tape). Participants will complete assessments before and after tape application. This pilot trial will inform future research interventions aiming to use the approach in different situations with pwMS (e.g., exercise).

DETAILED DESCRIPTION:
Research Plan

Participants The investigators will recruit and enroll 24 pwMS (12 per group) aged 18-55 years. This sample size is appropriate for pilot trials, and was not based on power analysis. The number of 12 per group is justified based on feasibility, gains in the precision about the mean and variance, and regulatory consideration. Related to gains in the precision, the gains are less pronounced after 12 participants. Recruitment will occur though advertisements in local newspapers (100-mile radius around Illinois campus) and posts on the Greater Illinois chapter of the National Multiple Sclerosis Society (NMSS) website. The investigators will further recruit using our participant's database that includes pwMS 40 years of age and older. The 24 persons will be randomly assigned in equal ratios through concealed allocation into either the intervention (i.e., Kinesio Tape - KTG; n=12) or control (i.e., Sham Tape - STG; n=12) conditions. The inclusion criteria are: clinically definitive diagnosis of MS; age between 18 and 55 years; relapse-free for the past 30 days and; ability to walk with or without assistive device (i.e., cane, but not walker/rollator). Participants further must be willing to complete in-person assessments in a university research setting. The investigators will exclude those who use wheelchair, crutches and walker or who have moderate cognitive impairment based on the modified Telephone Interview for Cognitive Status (i.e., moderate cognitive impairment, ≤ 12 points).

Main Outcomes

Balance. Balance will be objectively measured using a force platform (AccuSway, AMTI, Newton, MA, USA) which will be used to calculate the coordinates of the center of pressure (COP) during the standing test using three orthogonal forces and moments. Signals from the force plate will be sampled at 100HZ. Data analysis will then be performed using specific programs developed in MATLAB (Mathworks, Natick, MA, USA). Four classical time domain posturographic parameters will be calculated from the COP co-ordinates: mean deviation along the anterior-posterior (X) and medio-lateral (Y) axes, mean COP velocity along the anterior-posterior (VCOPX) and medio-lateral (VCOPY) axes. Participants will perform a total of four trials (i.e., two with eyes open and two with eyes closed) where they will be asked to stand on the force plate and maintain balance. The force plate will be set up 1.5 meters away from the wall. In the eyes open condition participants will be asked to focus at a dark disc (5cm in diameter) on the wall at the subject's eye level. Each trial will last one minute and participants will be given two minutes rest between trials. The order of the trial condition (eyes open or closed) will be randomized to prevent any order effect.

The Timed and up and Go test (TUG) will be used as a measure of functional mobility. The primary outcome of the TUG test is the total time (in seconds) taken to complete the test. The test will be set up on the basis of standardized descriptions that have been previously reported. Participants will be instructed to complete the course as safely and quickly as possible by standing up (without the help of hands), walking toward and around a cone/mark on the floor (approx. 10 feet), walking back to the chair, and then sitting down. If needed, participants will be allowed to use assistive devices while performing the task. Participants will be given 2 trials to complete the TUG test, and the average time across the 2 trials will be computed as the final score.

The Timed 25-foot Walk test (T25FW) will be used as a measure of walking speed. The primary outcome of the T25FW test is the total time (in seconds) taken to complete the test. Participants will be directed to one end of a clearly marked 25-foot course and will be instructed to walk 25 feet as quickly as possible, but within the limits of their safety. The time is calculated from the initiation of the instruction to start and ends when the participant has reached the 25-foot mark. If needed, participants may use assistive devices when performing the task. Participants will be given 2 trials to complete the T25FW test and the final score will be the average of the 2 completed trials.

The Six-minute Walking test (6MW) will be used as a measure of walking endurance. The primary outcome is the distance traveled at the end of 6 minutes with the use of a measuring wheel. The course is set up in a straight and clean hallway with at least 100-feet. Participants will be instructed to walk as quickly and safely as possible for 6 minutes making laps within 2 cones places 30 meters apart from each other. Participants will be allowed to use an assistive device if necessary and to rest when necessary. During the test participants will be followed by a second researcher who will walk to one side close enough for safety purposes. Only one trial is deemed to be appropriate and also helps avoiding fatigue.

The Six-spot Step test (SSST) will be used as a measure of lower-body coordination. The primary outcome of the SSST is the mean of the 4 trials in seconds. Participants complete the course as quickly as possible, while kicking the cones off of their labeled position with one foot, alternating between medial and lateral sides of the foot. Each participant completed the SSST four times: twice using their dominant foot, and twice using their non-dominant foot to kick the cones off of their demarcated position.

Experiment

Intervention Condition

Participants allocated into the Kinesio Tape Group (KTG) will receive a single time application of the kinesio tape flexible tape (Kinesio® Tex, Albuquerque, NM, USA) in the upper-body (i.e., back part of the trunk) and in the lower-body (i.e., legs and ankle) according to standardized procedures regarding tape application and participant skin preparation (https://kinesiotaping.com/how-to/). The tape is latex-free and wearable for weeks without causing skin irritation (i.e., hypoallergenic); and safe for populations ranging from pediatric to geriatric. The tape will be applied by a physical therapist with experience in tape application. Tape application will be conducted in a private room with complete structure for the procedure.

Control Condition

Participants allocated into the Sham Tape Group (STG) will receive a single time application of an inflexible tape (i.e., sham tape) in the same body segments as the intervention condition and applied by an experienced physical therapist. Tape application will be conducted in a private room with complete structure for the procedure.

Procedure

Recruitment ads/flyers will be created and posted. The study will be described as a non-invasive therapy approach to help improve balance, mobility and physical function. Interested persons will be asked to contact the Principal and co-Investigator (PI and Co-I) through telephone or email. Participant screening, contact, and enrollment will be undertaken over the telephone by a student involved in the project with the supervision of the Investigators. Those who are interested after the description will be screened for inclusion criteria. Participants meeting eligibility criteria who are interested in participating will be scheduled for a single test session for the provision of informed consent, demographic and anthropometric characteristics, and assessments of balance, mobility and physical function outcomes in the Department of Kinesiology and Physical Education. Participants will then be randomly assigned into either the KTG or STG group using concealed allocation. Participants will undertake the respective group-type tape application and will undergo the same assessment protocol as done for baseline.

Data-analysis

Dr. Zhang and Dr. Sebastião will be responsible for data analysis using SPSS software 24 version (SPSS Inc. Armonk, NY: IBM Corp.). The effect of the intervention will be examined using Condition × Time mixed-factor ANOVA with significance set a IP<.05. The partial eta-squared estimate for the interaction term from the ANOVA will inform power analyses for future Phase II trials, and the intra-correlation coefficient for test-retest reliability for the control group will inform the reliability estimate for the power analyses.

ELIGIBILITY:
Inclusion Criteria:

* clinically definitive diagnosis of MS
* aged 18 - 50 years
* relapse-free for the past 30 days and
* ability to walk with or without an assistive device (i.e., cane, but not walker/rollator).
* must be willing to complete in-person assessments at a university research setting

Exclusion Criteria:

* use wheelchair, crutches and walker
* have moderate cognitive impairment based on the modified Telephone Interview for Cognitive Status (i.e., moderate cognitive impairment, ≤ 12 points).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-25 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Static Balance Performance | 10minutes
  Center of Pressure (CoP) related measures collected from force plate
Timed and Up and Go | 6minutes
  a measure of functional mobility
Timed 25-foot Walk | 6minutes
  a measure of walking speed
Six-minute Walking Test | 10minutes
  a measure of walking endurance
Six-spot Step Test | 6minutes
  a measure of lower-body coordination
The Short Physical Performance Battery | 6minutes
  represent a recently validity measure of physical function in persons with MS

CONTACTS AND LOCATIONS:
Overall Officials: Emerson Sebastiao, PhD, Principal Investigator — Department of Kinesiology and Physical Education - Northern Illinois University
Locations (1):
- Department of Kinesiology and Physical Education. Northern Illinois University, DeKalb, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2008 Oct 25;372(9648):1502-17. doi: 10.1016/S0140-6736(08)61620-7. PMID 18970977
- [Background] Petzold A, Eikelenboom MJ, Keir G, Grant D, Lazeron RH, Polman CH, Uitdehaag BM, Thompson EJ, Giovannoni G. Axonal damage accumulates in the progressive phase of multiple sclerosis: three year follow up study. J Neurol Neurosurg Psychiatry. 2005 Feb;76(2):206-11. doi: 10.1136/jnnp.2004.043315. PMID 15654034
- [Background] Marrie RA, Yu N, Blanchard J, Leung S, Elliott L. The rising prevalence and changing age distribution of multiple sclerosis in Manitoba. Neurology. 2010 Feb 9;74(6):465-71. doi: 10.1212/WNL.0b013e3181cf6ec0. Epub 2010 Jan 13. PMID 20071664
- [Background] Bove R, Musallam A, Healy BC, Houtchens M, Glanz BI, Khoury S, Guttmann CR, De Jager PL, Chitnis T. No sex-specific difference in disease trajectory in multiple sclerosis patients before and after age 50. BMC Neurol. 2013 Jul 3;13:73. doi: 10.1186/1471-2377-13-73. PMID 23822612
- [Background] Dilorenzo T, Halper J, Picone MA. Reliability and validity of the multiple sclerosis quality of life inventory in older individuals. Disabil Rehabil. 2003 Aug 19;25(16):891-7. doi: 10.1080/0963828031000122195. PMID 12857582
- [Background] Finlayson M. Concerns about the future among older adults with multiple sclerosis. Am J Occup Ther. 2004 Jan-Feb;58(1):54-63. doi: 10.5014/ajot.58.1.54. PMID 14763636
- [Background] Finlayson M, Shevil E, Cho CC. Perceptions of cognitive symptoms among people aging with multiple sclerosis and their caregivers. Am J Occup Ther. 2009 Mar-Apr;63(2):151-9. doi: 10.5014/ajot.63.2.151. PMID 19432053
- [Background] Finlayson M, van Denend T. Experiencing the loss of mobility: perspectives of older adults with MS. Disabil Rehabil. 2003 Oct 21;25(20):1168-80. doi: 10.1080/09638280310001596180. PMID 14534060
- [Background] Jones KH, Ford DV, Jones PA, John A, Middleton RM, Lockhart-Jones H, Peng J, Osborne LA, Noble JG. How people with multiple sclerosis rate their quality of life: an EQ-5D survey via the UK MS register. PLoS One. 2013 Jun 11;8(6):e65640. doi: 10.1371/journal.pone.0065640. Print 2013. PMID 23776516
- [Background] Dalmonte J, Finlayson M, Helfrich C. In their own words: coping processes among women aging with multiple sclerosis. Occup Ther Health Care. 2004;17(3-4):115-37. doi: 10.1080/J003v17n03_08. PMID 23941225
- [Background] Shirani A, Zhao Y, Petkau J, Gustafson P, Karim ME, Evans C, Kingwell E, van der Kop ML, Oger J, Tremlett H. Multiple sclerosis in older adults: the clinical profile and impact of interferon Beta treatment. Biomed Res Int. 2015;2015:451912. doi: 10.1155/2015/451912. Epub 2015 Apr 1. PMID 25922836
- [Background] Alvarez-Alvarez S, Jose FG, Rodriguez-Fernandez AL, Gueita-Rodriguez J, Waller BJ. Effects of Kinesio(R) Tape in low back muscle fatigue: randomized, controlled, doubled-blinded clinical trial on healthy subjects. J Back Musculoskelet Rehabil. 2014;27(2):203-12. doi: 10.3233/BMR-130437. PMID 24284272
- [Background] Kim MK, Cha HG. The effects of ankle joint taping on gait and balance ability of healthy adults. J Phys Ther Sci. 2015 Sep;27(9):2913-4. doi: 10.1589/jpts.27.2913. Epub 2015 Sep 30. PMID 26504323
- [Background] Rojhani-Shirazi Z, Amirian S, Meftahi N. Effects of Ankle Kinesio Taping on Postural Control in Stroke Patients. J Stroke Cerebrovasc Dis. 2015 Nov;24(11):2565-71. doi: 10.1016/j.jstrokecerebrovasdis.2015.07.008. Epub 2015 Aug 29. PMID 26321149
- [Background] Nam CW, Lee JH, Cho SH. The effect of non-elastic taping on balance and gait function in patients with stroke. J Phys Ther Sci. 2015 Sep;27(9):2857-60. doi: 10.1589/jpts.27.2857. Epub 2015 Sep 30. PMID 26504310
- [Background] Kilbreath SL, Perkins S, Crosbie J, McConnell J. Gluteal taping improves hip extension during stance phase of walking following stroke. Aust J Physiother. 2006;52(1):53-6. doi: 10.1016/s0004-9514(06)70062-9. PMID 16515423
- [Background] Hsu YH, Chen WY, Lin HC, Wang WT, Shih YF. The effects of taping on scapular kinematics and muscle performance in baseball players with shoulder impingement syndrome. J Electromyogr Kinesiol. 2009 Dec;19(6):1092-9. doi: 10.1016/j.jelekin.2008.11.003. Epub 2009 Jan 14. PMID 19147374
- [Background] Cortesi M, Cattaneo D, Jonsdottir J. Effect of kinesio taping on standing balance in subjects with multiple sclerosis: A pilot study\m1. NeuroRehabilitation. 2011;28(4):365-72. doi: 10.3233/NRE-2011-0665. PMID 21725170
- [Background] Trojano M, Liguori M, Bosco Zimatore G, Bugarini R, Avolio C, Paolicelli D, Giuliani F, De Robertis F, Marrosu MG, Livrea P. Age-related disability in multiple sclerosis. Ann Neurol. 2002 Apr;51(4):475-80. doi: 10.1002/ana.10147. PMID 11921053
- [Background] Tintore M, Alexander M, Costello K, Duddy M, Jones DE, Law N, O'Neill G, Uccelli A, Weissert R, Wray S. The state of multiple sclerosis: current insight into the patient/health care provider relationship, treatment challenges, and satisfaction. Patient Prefer Adherence. 2016 Dec 22;11:33-45. doi: 10.2147/PPA.S115090. eCollection 2017. PMID 28053511
- [Background] Ford CC BR. Effects of aging on the disease course and management of multiple sclerosis. Sci. MS Manag. 2015;4:1-13
- [Background] Klaren RE, Sebastiao E, Chiu CY, Kinnett-Hopkins D, McAuley E, Motl RW. Levels and Rates of Physical Activity in Older Adults with Multiple Sclerosis. Aging Dis. 2016 May 27;7(3):278-84. doi: 10.14336/AD.2015.1025. eCollection 2016 May. PMID 27330842
- [Background] Thelen MD, Dauber JA, Stoneman PD. The clinical efficacy of kinesio tape for shoulder pain: a randomized, double-blinded, clinical trial. J Orthop Sports Phys Ther. 2008 Jul;38(7):389-95. doi: 10.2519/jospt.2008.2791. Epub 2008 May 29. PMID 18591761